CLINICAL TRIAL: NCT03334708
Title: Development of Biomarkers for the Early Detection, Surveillance and Monitoring of Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of Blood Based Biomarkers for Pancreas Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sheba Medical Center (Other Government); Weill Medical College of Cornell University (Other); Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: 17-527
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Pancreatic Diseases; Pancreatitis; Pancreatic Cyst
Keywords: 17-257
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Pancreatitis; Pancreatic Cyst | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be analyzed for various biomarkers. Initial biomarkers to be tested include proteins and proteases, functional DNA repair assays, exosomes, stromal elements, circular RNAs (cRNA) and circulating tumor DNA (ctDNA).
  Tissue will be utilized from already planned. Biopsy tissue is expected to be available for virtually all PDAC patients, occasionally for IPMN and cysts patients, rarely for pancreatitis and never for healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Locally Advanced or Metastatic Pancreatic Cancer Cohort: For patients with locally advanced or metastatic PDAC, blood will be collected pre-treatment initiation (baseline), after first chemotherapy cycle, every 8-12 weeks while under treatment to coincide with restaging CT scan and at time of disease progression.
  Interventions: Diagnostic Test: Blood Draw; Diagnostic Test: Tumor Tissue Collection
- Acute Benign Pancreatic Pathology Control Cohort: For patients with acute pancreatitis, blood specimens will be drawn at the time of acute pancreatitis and every 6-12 months thereafter
  Interventions: Diagnostic Test: Blood Draw; Diagnostic Test: Tumor Tissue Collection
- Chronic Benign Pancreatic Path,IPMC & Pancreatic Cyst Ctrl: For patients with chronic pancreatitis, IPMN, or cysts, blood specimens will be drawn every 6-12 months.
  Interventions: Diagnostic Test: Blood Draw; Diagnostic Test: Tumor Tissue Collection; Diagnostic Test: Cyst Fluid
- Healthy Control: For normal controls, blood specimens will be drawn once at study baseline.
  Interventions: Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Blood Draw — If clinically safe, up to approximately 50ml of blood will be drawn, not to exceed the following criteria:
  Patients and controls weighing 50kg or more
  * For draw amounts up to 50mL, there is no required hemoglobin threshold.
  * For amounts exceeding 50mL, patients who meet standard blood banking criteria (e.g., hemoglobin values within normal limits and minimum weight of 50kg) may give as much as a full unit of blood (500mL) at one time or in divided fractions over a 56 day/eight week period.
  Patients and controls weighing < 50kg
  * For patients whose hemoglobin is below normal limits but at least 7.0 gm/dL, no more than a total of 50 ml of blood or 5 ml/kg, whichever is less, may be collected per 56 day/eight week period, but no more than approximately 2 ml/kg of blood at any one time.
Diagnostic Test: Tumor Tissue Collection — Tumor tissue will be obtained by already planned biopsy, either at Memorial Sloan Kettering Cancer Center or elsewhere
  Groups: Acute Benign Pancreatic Pathology Control Cohort; Chronic Benign Pancreatic Path,IPMC & Pancreatic Cyst Ctrl; Locally Advanced or Metastatic Pancreatic Cancer Cohort
Diagnostic Test: Cyst Fluid — Cyst fluid will be obtained by already planned biopsy, either at Memorial Sloan Kettering Cancer Center or elsewhere
  Groups: Chronic Benign Pancreatic Path,IPMC & Pancreatic Cyst Ctrl

SUMMARY:
The purpose of this study is to develop a minimally invasive test to diagnose pancreatic cancer at early stages of disease and monitor response to treatment.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Advanced Pancreatic Cancer Cohort Inclusion Criteria

* Radiological, histological or cytological confirmed diagnosis of locally advanced or metastatic pancreatic adenocarcinoma by the enrolling institution
* Patient planning to receive systemic treatment
* Hemoglobin > 8
* ECOG performance status 0-2
* A minimum age of 18 years old
* Willing to undergo a tumor biopsy
* Willing to provide permission to obtain banked tumor tissue for analysis (previous biopsies or surgical material).

Cohort 2: Operable Pancreatic Cancer Cohort Inclusion Criteria

* Radiological, histological or cytological confirmed diagnosis of pancreatic adenocarcinoma by the enrolling institution
* Patient planned to undergo upfront resection
* No pre-operative systemic therapy nor chemoradiation therapy planned
* Hemoglobin > 8
* ECOG performance status 0-2
* A minimum age of 18 years old
* Willing to undergo a tumor biopsy
* Willing to provide permission to obtain banked tumor tissue for analysis (previous biopsies or surgical material).

Cohort 3: Acute Benign Pancreatic Pathology Control Inclusion Criteria

* Confirmed diagnosis of acute pancreatitis or other acute pancreatic pathology by the enrolling institution
* Hemoglobin > 8
* ECOG performance status 0-2
* A minimum age of 18 years old

Cohort 4: Chronic Benign Pancreatic Pathology Control Inclusion Criteria

* Confirmed diagnosis of chronic pancreatitis or other non-cystic chronic pancreatic pathology by the enrolling institution
* Hemoglobin > 8
* ECOG performance status 0-2
* A minimum age of 18 years old

Cohort 5: IPMN Control Inclusion Criteria

* Confirmed diagnosis of IPMN without high risk features by the enrolling institution
* A minimum age of 18 years old

Cohort 6: Pancreatic Cyst Control Inclusion Criteria

* Confirmed diagnosis of benign pancreatic cyst by the enrolling institution
* A minimum age of 18 years old

Cohort 7: Healthy Control Inclusion Criteria

* A minimum age of 18 years old

Exclusion Criteria:

Cohort 1: Advanced Pancreatic Cancer Cohort Exclusion Criteria

* Prior chemotherapy or radiation therapy for pancreatic cancer within the last 3 months in the localized setting
* Active second malignancy, unless low grade malignancy
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 2: Operable Pancreatic Cancer Cohort Exclusion Criteria

* Neoadjuvant chemotherapy or radiation therapy is planned
* Active second malignancy, unless low grade malignancy
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 3: Acute Benign Pancreatic Pathology Control Exclusion Criteria

* Active or prior malignancy, except prior non-melanoma skin cancer
* Proven to be a carrier of a cancer susceptibility gene or family history concerning for genetic predisposition to cancer
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 4: Chronic Benign Pancreatic Pathology Control Exclusion Criteria

* Active or prior malignancy, except prior non-melanoma skin cancer
* Proven to be a carrier of a cancer susceptibility gene or family history concerning for genetic predisposition to cancer
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 5: IPMN Control Exclusion Criteria

* IPMN with high risk features or planned resection
* Active or prior malignancy, except prior non-melanoma skin cancer
* Proven to be a carrier of a cancer susceptibility gene or family history concerning for genetic predisposition to cancer
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 6: Pancreatic Cyst Control Exclusion Criteria

* Active or prior malignancy, except prior non-melanoma skin cancer
* Proven to be a carrier of a cancer susceptibility gene or family history concerning for genetic predisposition to cancer
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Cohort 7: Healthy Control Exclusion Criteria

* Active or prior malignancy, except prior non-melanoma skin cancer
* Proven to be a carrier of a cancer susceptibility gene or family history concerning for genetic predisposition to cancer
* Any medical or psychiatric condition that may interfere with ability to comply with protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects in the PDAC and benign pancreatic disease cohorts will be identified by a member of the patient's treatment team, the principal investigator, or research team at participating institutions. If the investigator is a member of the treatment team, s/he will screen their patients' medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. The investigator will use information provided by the patient and/or medical record to confirm that the patient is eligible and contact the patient regarding study enrollment. Healthy controls will be recruited from patients from outpatient primary care clinics at non-MSK sites and volunteers from which may include the staffs members at collaborating sites.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in biomarkers to determine sensitivity and specificity of the assay to diagnose early stage pancreatic cancer | 4 years

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Cold Springs Harbor Laboratory (Specimen Analysis), Cold Spring Harbor, New York
  - Memorial Sloan Kettering Cancer Center @ Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - New York University, New York, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York
- Israel (3):
  - Sha'are Zedek Medical Center, Jerusalem
  - Weizmann Institute of Science, Rehovot
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org